CLINICAL TRIAL: NCT00397800
Title: Safety and Efficacy of Sequential Treatment With a Combination of Rituximab, Fludarabine and Cyclophosphamide Followed by Zevalin (Rituximab and Y-Ibritumomab Tiuxetan) - A Phase I/II Study for Treatment of Patients With Relapsed Indolent and Transformed CD20-Positive B-Cell Non-Hodgkin's-Lymphoma Ineligible for High-Dose Chemo(Radio)Therapy Supported by Autologous Peripheral Blood Stem-Cells
Brief Title: Rituximab, Fludarabine, Cyclophosphamide, and Yttrium Y 90 Ibritumomab Tiuxetan in Treating Patients With Relapsed B-Cell Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000515982; KRDI-TUM-R-F-015-V-0030-I; EU-20633
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; Waldenstrom macroglobulinemia; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Waldenstrom Macroglobulinemia; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Rituximab; Cyclophosphamide; fludarabine phosphate; ibritumomab tiuxetan

INTERVENTIONS:
Biological: rituximab
Drug: cyclophosphamide
Drug: fludarabine phosphate
Radiation: yttrium Y 90 ibritumomab tiuxetan

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy, such as fludarabine and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Radiolabeled monoclonal antibodies, such as yttrium Y 90 ibritumomab tiuxetan, can find cancer cells and carry cancer-killing substances to them without harming normal cells. Giving rituximab and chemotherapy together with yttrium Y 90 ibritumomab tiuxetan may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of yttrium Y 90 ibritumomab tiuxetan when given together with rituximab, fludarabine, and cyclophosphamide and to see how well they work in treating patients with relapsed B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the dose-limiting toxicity and maximum tolerated dose of rituximab and yttrium Y 90 (^90Y) ibritumomab tiuxetan when administered with rituximab as radioimmunotherapy after rituximab, fludarabine, and cyclophosphamide in patients with relapsed indolent, mantle cell, or transformed CD20-positive B-cell non-Hodgkin's lymphoma.

Secondary

* Determine the overall survival in patients treated with this regimen.
* Determine time to progression and event-free survival in patients treated with this regimen.
* Determine partial and complete response rates in patients treated with this regimen.
* Determine time to maximal response in patients treated with this regimen.
* Determine response duration in patients treated with this regimen.
* Determine the feasibility of additional antineoplastic treatment following disease relapse after treatment with rituximab and ^90Y ibritumomab tiuxetan in these patients.

OUTLINE: This is a prospective, nonrandomized, multicenter, phase I dose-escalation study of yttrium Y 90 (^90Y) ibritumomab tiuxetan followed by a phase II open-label study.

* Phase I:

  * Chemoimmunotherapy: Patients receive rituximab IV on day 1 and fludarabine IV over 30 minutes and cyclophosphamide IV over 60 minutes on days 1-3. Treatment repeats every 4 weeks for up to 3 courses in the absence of disease progression. Four weeks after the first day of the last chemoimmunotherapy course, patients receive 1 dose of rituximab IV alone. Patients with disease progression are removed from the study. Patients with stable disease proceed to radioimmunotherapy 8-12 weeks after the first day of the last chemoimmunotherapy course.
  * Radioimmunotherapy: Patients receive rituximab IV and an imaging dose of indium In III ibritumomab tiuxetan IV over 10 minutes on day 1. Patients then undergo imaging. If dosimetry is acceptable, patients receive rituximab IV and ^90Y ibritumomab tiuxetan IV over 10 minutes on day 8.

Cohorts of 3-6 patients receive escalating doses of ^90Y ibritumomab tiuxetan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive chemoimmunotherapy and radioimmunotherapy as in phase I, at the MTD determined in phase I.

Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 2 years.

PROJECTED ACCRUAL: A total of 12 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed CD20-positive B-cell non-Hodgkin's lymphoma (NHL), including any of the following subtypes:

  * Indolent NHL, including any of the following:

    * Follicular
    * Lymphoplasmacytoid
    * Marginal zone
  * Mantle cell NHL
  * Transformed B-cell NHL
* In at least first relapse with an indication for systemic antineoplastic treatment, as defined by the following:

  * Local or constitutional (B-) symptoms
  * Hypersplenism due to splenic involvement
  * Bulky disease (> 7.5 cm in diameter)
  * Impending medical problems derived from rapid disease progression within the past 6 months, as defined by an observed or anticipated > 50% increase in the sum of the areas calculated from multiplying the greatest perpendicular diameters of each lesion
* Measurable lesions of lymphoma infiltration
* Medically ineligible for high-dose treatment followed by autologous stem cell support
* Adequate bone marrow cellularity (> 15% of marrow area covered by hematopoiesis)
* No CNS, leptomeningeal, spinal cord, or testes lymphoma involvement
* No lymphoma lesion mandating emergency radiotherapy
* No clinical, cytological, cytogenetic, or histopathologic indication of myelodysplastic syndrome
* If there is bone marrow infiltration detected prior to chemoimmunotherapy, patient must undergo a repeat bone marrow biopsy prior to planned treatment with radioimmunotherapy to verify the level of bone marrow infiltration is < 25%

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* Absolute neutrophil count > 1,500/mm³
* Platelet count > 150,000/mm³
* Hemoglobin > 9 g/dL
* Creatinine < 1.5 times upper limit of normal (ULN)
* Bilirubin < 2 times ULN
* ALT and AST < 2 times ULN
* Albumin > 2.5 g/dL
* INR < 1.5
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 12 months after completion of study treatment
* No concurrent severe and/or uncontrolled medical disease that would preclude study compliance, including any of the following:

  * Uncontrolled diabetes
  * Congestive heart failure
  * Chronic renal disease
  * Active uncontrolled infection
* No bleeding risks or disorders, including any of the following:

  * CNS abnormalities suggesting an increased susceptibility for hemorrhage, including recent history of stroke as demonstrated by cranial contrast-enhanced CT scan
  * Severe arrhythmia or uncontrolled hypertension
  * Myocardial infarction within the past 6 months
  * Diabetic retinopathy with history of symptomatic hemorrhage
  * Known and potentially active gastrointestinal bleeding foci
  * Concurrent anticoagulant medication that must be continued even with platelet count < 20,000/mm³ (e.g., following mitral valve replacement, anti-phospholipid syndrome, or recurrent venous thromboembolism)
  * Other congenital or acquired hemorrhagic diatheses
* No ongoing autoimmune hemolytic anemia
* No known presence of anti-murine antibody reactivity
* No known hypersensitivity to murine or chimeric antibodies or proteins
* No known HIV infection
* No psychiatric illness that would preclude study requirements
* No other malignant disorder within the past 10 years except basal cell carcinoma of the skin or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* No more than 4 prior systemic anti-lymphoma regimens (including single-agent rituximab)
* At least 2 months since prior systemic anti-lymphoma treatment (including single-agent rituximab)
* No prior radioimmunotherapy
* No prior autologous or allogeneic hematopoietic stem cell transplantation
* No prior treatment with purine analogues that has not resulted in remission for > 1 year
* No prior anti-CD20 radioimmunoconjugate therapy
* More than 5 years since prior radiotherapy to extensive fields covering lymph node regions on both sides of the diaphragm or > 50% of the spinal column
* More than 4 weeks since prior surgery
* No concurrent oral anticoagulant therapy

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2005-06; Primary Completion 2008-05 (Actual); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity

SECONDARY OUTCOMES:
Response
Survival

CONTACTS AND LOCATIONS:
Overall Officials: Christian Peschel, MD, Study Chair — Technical University of Munich
Locations (12):
- Germany (12):
  - Medizinische Klinik, Klinikum Augsburg, Augsburg
  - Medizinische Klinik III - Universitaetsklinikum Erlangen, Erlangen
  - Universitaetsklinikum Goettingen, Göttingen
  - Universitaetsklinikum Schleswig-Holstein - Campus Luebeck, Lübeck
  - Universitaetsklinkum Magdeburg der Otto-von-Guericke-Universitaet Magdeburg, Magdeburg
  - Universitatsklinik Mainz, Mainz
  - LMU-Klinikum Grosshadern, Munich
  - Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich
  - Klinikum der Universitaet Regensburg, Regensburg
  - Universitaetsklinikum Tuebingen, Tübingen
  - Comprehensive Cancer Center Ulm at Universitaetsklinikum Ulm, Ulm
  - Medizinische Klinik und Poliklinik II - Universitaetsklinikum Wuerzburg, Würzburg